CLINICAL TRIAL: NCT07229326
Title: POSITIVE OUTCOMES: Driving up the Quality of HIV Outpatient Care Through the Routine Implementation of a PROM to Promote Patient-centredness
Brief Title: POSITIVE OUTCOMES: Improving Quality
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IN-UK-985-6892
Record Dates: First submitted 2025-09-24; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: Patient-Reported Outcomes; Implementation; Patient-Reported Outcome Measures; Quality Improvement; Person-Centred Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- People Living with HIV
  Interventions: Other: POSITIVE OUTCOMES

INTERVENTIONS:
Other: POSITIVE OUTCOMES — POSITIVE OUTCOMES is a validated patient-reported outcome measure

SUMMARY:
People Living with HIV (PLWH) in the UK have a high burden of mental health, social and spiritual concerns, physical symptoms, and poorer health-related quality of life than the general population. PLWH feel that routine clinical appointments do not routinely address the things that matter to them, with implications for their engagement and outcomes of treatment and care. Contrastingly, good psychosocial care and communication with HIV professionals are associated with improvements in clinical outcomes, adherence and retention in care. Although HIV service structures, processes and outputs are routinely audited, it is person-centred patient-reported outcomes that define quality care. We have established a stakeholder project team, conducted community consultation and undertaken careful research-led development of a PROM for PLWH (called "POSITIVE OUTCOMES". This PROM has been developed in 2 European countries and validated in 5 European countries, using best scientific principles of psychometrics. We have established face and content validity, conducted cognitive interviews, and demonstrated validity and reliability in a sample of N=1,705 PLWH who completed at least 2 data points (manuscript in preparation). This was conducted alongside a national consultation to develop the new iteration of HIV care standards that includes a standard on "person-centred care" https://www.bhiva.org/file/KrfaFqLZRlBhg/BHIVA-Standards-of-Care-2018.pdf.

To meet the requirements in delivering and auditing person-centred care within those standards, we need to answer the following questions:

* What are optimal methods for routine implementation of the PROM from the perspectives of stakeholders
* What are locally-relevant components of a Decision Support Tool to provide clinicians with appropriate evidence-based clinical responses to patient PROM scores
* What is an implementable Quality Improvement Programme to improve person-centred outcomes, informing (inter)national roll out with existing registry data?

The aim of this proposal is to develop a five-site demonstration patient-centred quality improvement programme determining feasibility, optimal implementation methods and data usage, and to deliver a framework for (inter)national adoption.

The objectives are:

* To develop a quality improvement team within each of our three demonstration sites and identify site-specific challenges and potential solutions (including IT) for PROM implementation.
* To develop an evidence-based Decision Support Tool (DST) specifying clinical responses to real-time PROM data from PLWH that are feasible within local resources, a PROM training programme for clinicians and a PLWH "mentor" for patients in each site
* Hold a quality improvement launch meeting to train on POSITIVE OUTCOMES and DST implementation.
* Implement the Positive Outcomes PROM in three demonstration sites
* Test impact on outcomes using annual quality improvement cycles at facility level Determine stakeholder (PLWH, clinician) views on the quality improvement mechanisms, impact and areas for further refinement.
* Develop and disseminate a national manual on implementation of the POSITIVE OUTCOMES quality improvement programme.

The project is working with 5 clinics across the UK and the US:

* King's College Hospital NHS Foundation Trust (London, UK)
* Chelsea and Westminster Hospital (London, UK)
* Brighton and Sussex University Hospitals NHS Trust (Brighton, UK)
* HOWARD BROWN Health Clinic (Chicago, US)
* CAN SUPPORT Community Health Center (Miami, US)

The observational model for the project is a quality improvement programme.

ELIGIBILITY:
Inclusion Criteria:

* adult (aged at least 18 years) attending outpatient HIV care at one of the UK recruitment sites
* able to consent to participate in the study
* able to communicate in English or a language provided by NHS translation services
* purposively sampled by age, gender, ethnicity, sexual orientation, and time since HIV diagnosis

Exclusion Criteria:

* Aged under 18
* not attending care at one of the recruitment sites
* not able to consent to participate in the study
* speaks a language not available through NHS translation services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV who regularly attend one of the five study clinics.
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Stakeholder views | 6-24 months
  Determine stakeholder views through longitudinal qualitative in-depth interviews with people living with HIV who have completed the POSITIVE OUTCOMES PROM. 4-6 weeks after each interview, the participant's case notes will be reviewed alongside the completed PROM to examine what documented actions have been made in response to symptoms and concerns raised using the PROM.
  Additionally, approximately 15 clinicians and staff from each UK site will be recruited to participate in focus groups 6 months before the end of the 2 year implementation period. Topic guides will address the PROM content, timing and method of completion, data sharing, use of data in clinical encounters, response of clinical team to the PROM data, perceived impact of using the PROM and the perceived mechanisms of action for any impact. We will also seek to elicit any suggested improvements for the programme and recommendations for the national roll-out manual.

REFERENCES:
- [Background] Harding R, Clucas C, Lampe FC, Date HL, Fisher M, Johnson M, Edwards S, Anderson J, Sherr L. What factors are associated with patient self-reported health status among HIV outpatients? A multi-centre UK study of biomedical and psychosocial factors. AIDS Care. 2012;24(8):963-71. doi: 10.1080/09540121.2012.668175. Epub 2012 Apr 23. PMID 22519889
- [Background] Bristowe K, Clift P, James R, Josh J, Platt M, Whetham J, Nixon E, Post FA, McQuillan K, Ni Cheallaigh C, Murtagh F, Anderson J, Sullivan AK, Harding R. Towards person-centred care for people living with HIV: what core outcomes matter, and how might we assess them? A cross-national multi-centre qualitative study with key stakeholders. HIV Med. 2019 Sep;20(8):542-554. doi: 10.1111/hiv.12758. Epub 2019 Jun 4. PMID 31162817
- [Background] Bristowe K, Murtagh FEM, Clift P, James R, Josh J, Platt M, Whetham J, Nixon E, Post FA, McQuillan K, Cheallaigh CN, Kall M, Anderson J, Sullivan AK, Harding R. The development and cognitive testing of the positive outcomes HIV PROM: a brief novel patient-reported outcome measure for adults living with HIV. Health Qual Life Outcomes. 2020 Jul 6;18(1):214. doi: 10.1186/s12955-020-01462-5. PMID 32631444
- [Background] Harding R, Jones CI, Bremner S, Bristowe K, West B, Siegert RJ, O'Brien KK, Whetham J; EMERGE Consortium, Horizon 2020. Positive Outcomes: Validity, reliability and responsiveness of a novel person-centred outcome measure for people with HIV. HIV Med. 2022 Jul;23(6):673-683. doi: 10.1111/hiv.13224. Epub 2022 Jan 11. PMID 35014143
- See also: Project Website — https://www.kcl.ac.uk/research/positive-outcomes-improving-quality